CLINICAL TRIAL: NCT00925158
Title: Non-randomized Clinical Trial for Evaluation of the Dissector Assisted Malar Elevation in Videoendoscopic Rhytidoplasty.
Brief Title: Dissector Assisted Malar Elevation for Rhytidoplasty
Acronym: DAME
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, LYDIA MASAKO FERREIRA, MD, PhD, Federal University of São Paulo
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: CEP-UNIFESP 1515/07
Record Dates: First submitted 2009-06-18; First posted 2009-06-19 (Estimated); Last update posted 2012-07-24 (Estimated); Status verified 2012-07

CONDITIONS: Aging; Premature Aging
Keywords: Rhytidoplasty; Video-Assisted Surgery; Surgical instruments; Dissection; Innovative therapies; Face; Aging; Premature aging; Rejuvenation
MeSH Terms: conditions — Aging, Premature; Facies | interventions — Rejuvenation; Rhytidoplasty; Video-Assisted Surgery

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Surgical instrument (DAME) (Experimental): Surgical dissector instrument created to malar elevation.
  Interventions: Procedure: Dissector Assisted Malar Elevation

INTERVENTIONS:
Procedure: Dissector Assisted Malar Elevation — Malar dissector - Surgical instrument for video endoscopic rhytidoplasty.
  Other Names: Face; Rejuvenation; Rhytidoplasty; Video-Assisted Surgery; Malar fat pad; Image Processing; Computer-Assisted; Malar dissector

SUMMARY:
BACKGROUND: Endoscopy was first used in plastic surgery for the treatment of frontal rhytides. This minimally invasive approach allows the treatment of frontal wrinkles using a practical procedure that does not directly interfere with the frontalis muscle, acting only on its antagonists.

It is also possible to treat the middle third of the face, but these evolutions depends on special surgical instruments. Videoendoscopic approach in rhytidoplasty have been improved by new devices and surgical instruments.

The mid third of the face can be treated in different ways. Zygomatic projection can be achieved by the use of the Dissector Assisted Malar Elevation (DAME) procedure.

AIM: Evaluate the zygomatic projection achieved by DAME in videoendoscopic rhytidoplasties.

METHODS: 30 non-white female patients, 30 to 59 years old, will be submitted to videoendoscopic rhytidoplasty with malar elevation by the DAME. Pre- and post-operative facial appearance will be evaluated by digital photogrammetry.

DETAILED DESCRIPTION:
THE NEW SURGICAL INSTRUMENT:

The dissector developed by the authors is a stainless steel instrument, 20 cm in length, 1 cm in diameter, with a cylindrical handle, and an articulated section 3 cm in length and 1cm in diameter at the distal end. When the most proximal end of the handle is rotated, the articulated section provides for angulation or articulation of the distal end portion with respect to the longitudinal axis of the instrument that is similar to the movements of a distal phalanx of a finger.

SURGICAL TECHNIQUE:

1. Frontal Region: An incision line, 2 cm long, in the median sagittal plane and 1 cm from the hairline; an incision line, 2 cm long, parallel and 4 cm from the sagittal line, to the right and left sides;
2. Temporal Region: An incision line, 3 cm long, 3 cm from the hairline, perpendicular to and bisected by a line traced from the margin of the nasal wing, passing by the lateral palpebral commissure and extending in the posterior direction, bilaterally.

Following, the hair was gathered into bundles to allow access to the skin markings, and held by latex rings, which were obtained by cross-sectional cuts through fingers of sterile latex surgical gloves.

Skin antisepsis was performed with 0.2% aqueous chlorhexidine, followed by the placement of sterile surgical drapes, and retracing of the sagittal, parasagittal and temporal incision lines (described above) with methylene blue.

The right temporal incision was performed on the marked area, cutting through the skin and superficial temporal fascia, and exposing the deep temporal fascia. Following, the undermining of the temporal region surrounding the incision was carried out in the interfascial plane, under direct vision, to prepare the optical cavity. The dissection proceeded to the orbital and zygomatic regions, under endoscopic vision, using a rigid endoscope (Karl Storz, model 7230 BWA) 18cm in length, 4mm in diameter and with a 30-degree angle. The dissection continued until the medial zygomatic-temporal vein (also known as sentinel vein) was reached; a xenon light source (Karl Storz, model 20131501) was used to illuminate the optical cavity.

The zygomatic-temporal vein was previously cauterized with an endoscopic grasper (Karl Storz, model 50232 GG) and incised with scissors (Karl Storz, model 50231 GW) to allow dissection toward the lateral orbital rim. In this region, after passing the lateral palpebral ligament, the undermining ?) deepened, becoming subperiosteal on the zygomatic bone. The subperiosteal undermining ?) progressed along the whole inferior orbital rim up to its most medial portion, superior to the infraorbital nerve, to completely release the inferior orbital rim under endoscopic vision with the aid of an elevator (Karl Storz, model 50205s).

Using the same surgical instrumentation, a subcutaneous tunnel was created from the temporal incision towards the middle third of the face until the inferolateral limit of the orbicularis oculi muscle was reached. From this point, a blunt dissection of the malar fat pad was performed with the use of a dissector instrument, which had been developed for this purpose, as described by the author in 2004 and published in 2006. After blunt dissection, the malar fat pad was projected in the antero-superior direction by means of a suture in the zygomatic projection to restore the zygomatic contour and the anterior projection of the middle third of the face. The above procedures were then repeated on the contralateral hemiface.

The procedure was continued with the frontal incisions, which were previously described, by cutting through the skin to the periosteum (fig. 2). A subperiosteal dissection of the entire frontal region was performed to a distance of 1 cm above the eyebrow.

Under endoscopic vision, the dissection proceeded to the glabella, where the periosteum was incised with a sharp dissector to expose the bone insertions of the procerus, corrugator and depressor supercilii muscles. A thin dissector and an endoscopic grasper with a diathermy cable (unipolar high-frequency cord, model 26002 M, Karl Storz) were used in the myotomy and partial myectomy of these muscles. This periosteotomy started at the glabella region, and continued transversally toward the lateral end of the eyebrow in both sides, passing by the supratrochlear nerve, and reaching the supraorbital nerve, where it was interrupted to be continued in a latero-medial direction in the next surgical step.

The frontal and temporal undermining were united by the incision of the temporal ligament with a sharp dissector, exposing its most inferior portion, where the Hakme ligament is located. This ligament was incised with endoscopic scissors; this maneuver simultaneously released the lateral margin of the detached periosteum. At this level, the periosteotomy continues marginal to the orbital rim in a lateral-medial direction to the supraorbital nerve, which was identified and isolated. All fibrous adhesions of the body and tail of the eyebrow found in this path were dissected using a sharp dissector until the fibers of the palpebral portion of the orbicularis oculi muscle were reached at this level, completing the horizontal periosteotomy in its entire extension, the treatment of structures, and the undermining of the periorbital, frontal and temporal regions.

For the patients in the fixation group, the fixation points of the frontal flap were determined as the intersection point between the parasagittal line that passes through the transition of the lateral third with the two medial thirds of the eyebrow and the hairline. This point was called FEP (flap elevation point).

After attaching one end of a 2-0 nylon monofilament thread to the deep temporal fascia, a Casagrande needle was inserted at the FEP, penetrating the skin and periosteum, and transfixing the point. Following, the needle was directed to the deep temporal fascia at the fixation level. At this level, the other end of the nylon thread was passed through the hole of the Casagrande needle. The needle was pulled back to the FEP and, at this point, the periosteum was transfixed from depth to surface, up to the deep dermis. Then, the needle was returned to the depth, to a point located 0.5 cm medially, in order to fix the flap at the FEP level. The needle was directed to the sagittal incision, where once more it penetrated in the periosteum from depth to surface, externalizing the nylon thread. The same procedure was performed on the contralateral side. The two free ends of both nylon threads were tied together with a surgical knot at their emergence point along the sagittal plane with enough traction to elevate and fix the eyebrow to a position immediately superior to the superior orbital rim.

The incisions were closed with 4-0 monofilament nylon suture on a 2cm triangular needle; the detached site was drained by a closed vacuum system, with a drain tube (size 10) fixed to the sagittal incision and maintained for 48 hours. The skin was cleansed with 0.9% saline solution, tincture of benzoin was applied, and self-adhesive microporous tape (Micropore) was used and maintained for 7 days.

PHOTOGRAPHIC STANDARDIZATION:

Photographs were taken from all patients in a standardized manner, with respect to the equipment, camera positioning, lighting conditions, and positioning of the cephalic segment in relation to the Frankfurt plane. Photographs were taken in frontal view preoperatively and at 12 months postoperatively.

DIGITAL PHOTOGRAMMETRY:

Image analysis was done on a personal computer using the UTHSCSA ImageTool Version 3.0 software for Windows.

Digital photogrammetric measurements were made based on the anthropometric landmarks Endocathion (EN), which corresponds to the medial palpebral commissure, and Exocathion (EX), which corresponds to the lateral palpebral commissure.22-24 The distance between the EN-right and EN-left points (EN-EN distance) was measured. The length of a paramedian vertical line, connecting the intersection of the lateral extension of the EN-EN line with the EX point to the intersection of the EN-EN line with the outer margin of the eyebrow, which was denominated EB (eyebrow) or distance EX-EB, was also measured.

Based on the photographs, the Brow Position Index (BPI) was calculated for both the right (BPIR) and left (BPIL) sides. The BPI was defined as the ratio between the EN-EN (in pixels) and EX-EB (in pixels) distances multiplied by 100. Following, the difference (delta), in absolute value, between the preoperative BPI (BPI-pre) and 12month postoperative BPI (BPI-post) was calculated for both sides.

ELIGIBILITY:
Inclusion Criteria:

* white and non-white
* premature facial aging

Exclusion Criteria:

* diabetes
* arterial hypertension
* any previous facial aesthetic therapy

Ages: 30 Years to 59 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2007-12; Primary Completion 2012-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Digital photogrammetry | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Lydia M Ferreira, M.D., PhD., Principal Investigator — Plastic Surgery Division - Professor. Surgery Department - Chairwoman and Head.
Locations (1):
- Hospital São Paulo - UNIFESP, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Ferreira LM, Horibe EK. Understanding the finger-assisted malar elevation technique in face lift. Plast Reconstr Surg. 2006 Sep;118(3):731-40. doi: 10.1097/01.prs.0000233050.10568.66. PMID 16932185